CLINICAL TRIAL: NCT04880798
Title: Effect of Thyrotropin Level on Iodine Uptake: a Prospective 124I PET/CT Study in Metastatic Differentiated Thyroid Cancer
Brief Title: Effect of Thyrotropin Level on Iodine Uptake in Metastatic Differentiated Thyroid Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yansong Lin, Prof, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-BCH-124I
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Differentiated Thyroid Cancer
Keywords: differentiated thyroid cancer; pulmonary metastases; bone metastases; thyrotropin; thyroid stimulating hormone; 124I PET/CT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 124I PET/CT (Experimental): All eligible patients will be allocated to this arm (single-arm study).
  Interventions: Diagnostic Test: 124I PET/CT

INTERVENTIONS:
Diagnostic Test: 124I PET/CT — The first 124I PET/CT was prepared with endogenous thyrotropin 30±10 μIU/mL, and the second 124I PET/CT was prepared with endogenous thyrotropin >100 μIU/mL. The RAI-avidity of the metastases was assessed twice along with the levothyroxine withdrawal by 124I PET/CT scans.

SUMMARY:
Distant metastases is the leading cause of differentiated thyroid cancer-related death. Radioactive iodine (RAI) treatment is the most effective therapy for RAI-avid metastatic differentiated thyroid cancer (DTC). It is well known that the efficacy of RAI therapy is depend on the sodium-iodide symporter protein, which can be synthesized by elevated thyrotropin stimulation. Therefore, thyrotropin stimulation before RAI treatment to ensure sufficient uptake of RAI has been a long-established procedure. According to some observational studies, thyrotropin of 25-30 μIU/mL has been adopted as the standard care protocol. However, whether thyrotropin of 25-30 μIU/mL is enough to stimulate iodine uptake in metastatic lesions remains unknown. In this study, the investigators aim to address the effect of thyrotropin on iodine uptake in metastatic DTC during levothyroxine withdrawal by two times 124I PET/CT scans on different endogenous thyrotropin levels.

DETAILED DESCRIPTION:
It is estimated that 10 patients who met the study criteria will be enrolled. All patients underwent twice 124I PET/CT scans in Beijing Cancer Hospital. The first 124I PET/CT was prepared with endogenous thyrotropin 30±10 μIU/mL, the second 124I PET/CT was prepared with endogenous thyrotropin >100 μIU/mL. The RAI-avidity of the metastases was assessed twice along with the levothyroxine withdrawal by 124I PET/CT scans.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent total thyroidectomy.
2. Patients were diagnosed with differentiated thyroid cancer by postoperative pathological examination.
3. Distant metastases confirmed by CT etc.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Significant hepatic or renal dysfunction;
3. Unable to lie flat, still or tolerate a PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of thyrotropin level on iodine uptake in metastatic DTC lesions on twice 124I PET/CT. | 1 month
  SUV metrics of RAI-avid metastatic DTC lesions on twice 124I PET/CT.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing